CLINICAL TRIAL: NCT07008742
Title: Feasibility Study of Tissue and Blood Collection in Oncogene-addicted and Neoadjuvantly Treated Non Small Cell Lung Cancer
Acronym: FeStival
Status: Recruiting | Type: Observational
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: Francis Crick Institute (Other); University of Cambridge (Other); Royal Brompton & Harefield NHS Foundation Trust (Other); Institute of Cancer Research, United Kingdom (Other)
Responsible Party: Sponsor
Other Study IDs: CCR5952; 336531 (Other: Integrated Research Application System (IRAS)); 24/LO/0791 (Other: Research Ethics Committee)
Record Dates: First submitted 2025-05-15; First posted 2025-06-06 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Oncogene-addicted Non Small Cell Lung Cancer; Early-stage Operable Non Small Cell Lung Cancer; Non Small Cell Lung Cancer; Metastatic Non Small Cell Lung Cancer; Locally Advanced NSCLC - Non-Small Cell Lung Cancer; Stage 2/3 Operable Non Small Cell Lung Cancer
Keywords: tissue; blood; feasibility study
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Archival tissue, fresh surgical tissue, blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Cohort 1A: Treatment naïve, oncogene-addicted NSCLC
- Cohort 1B: Pre-treated, oncogene-addicted NSCLC, received prior targeted therapy
- Cohort 1C: Pre-treated, oncogene-addicted NSCLC, no prior targeted therapy (can have received chemotherapy/CPI/chemo-CPI)
- Cohort 2: Early-stage operable NSCLC undergoing neoadjuvant CPI therapy

SUMMARY:
This study aims to determine if it is feasible to collect samples of blood and viable lung cancer tissue in patients with either:

* Stage IV mutation-driven NSCLC
* Stage II-III NSCLC undergoing neoadjuvant immunotherapy prior to surgery

Viable tissue has been defined by the collaborating pathology department as the presence of viable tumour cells, in accordance with recommendations from the International Association or the Study of Lung Cancer.

In patients with stage IV NSCLC, obtaining adequate samples of viable tissue for advanced testing can be challenging, as sites of cancer that are accessible by biopsy are often small, and contain few viable cancer cells. If obtained, however, viable blood and tissue specimens can be utilised for genetic and other analyses aimed at identifying cancer markers that may offer prognostic information, or that may potentially lead to development of therapies that target these markers in the future.

In patients with stage II-III NSCLC, the use of immunotherapy prior to surgery has been shown to affect the proportion of viable tumour tissue at the time of surgery, although this needs to be further studied. There is a need to better understand the genetic basis of these tumours to improve response rates to immunotherapy prior to surgery.

The study will be open for four years in total. The first three years will consist of recruitment and participant follow up, and the fourth year will consist of follow up only. Data analysis will occur in the fifth year when the study is closed.

DETAILED DESCRIPTION:
Rationale Benchmarking the proportion of patients who are able to provide paired samples of blood and viable tumour tissue is important in oncogene-addicted metastatic NSCLC patients as investigators have now entered the era of genotype-guided post-progression targeted therapies. In the early-stage operable NSCLC context, benchmarking the feasibility of paired samples is of interest as neoadjuvant CPI-based therapy has recently emerged as a new standard of care strategy.

As such, investigators have defined the following cohorts within our study:

Cohort 1: Oncogene-addicted NSCLC, due to commence new line of targeted therapy

* Sub-cohort 1A: treatment naïve, oncogene-addicted NSCLC
* Sub-cohort 1B: pre-treated, oncogene-addicted NSCLC, received prior targeted therapy
* Sub-cohort 1C: pre-treated, oncogene-addicted NSCLC, no prior targeted therapy (can have received chemotherapy/CPI/chemo-CPI) Cohort 2: Early-stage operable NSCLC undergoing neoadjuvant CPI therapy

Primary aim

To estimate the feasibility of collecting paired samples of blood and viable tissue in patients with:

* Oncogene-addicted metastatic NSCLC commencing new line of targeted therapy at progression (Cohort 1), and
* Early-stage operable NSCLC undergoing neoadjuvant CPI-based therapy (Cohort 2) Viable tissue is defined by the presence of viable tumour cells. Viable tumour cells are defined by those with well-preserved architectural and cytological features, in line with the latest recommendation from the International Association for the Study of Lung Cancer (IASLC), evaluated by a specialist pulmonary pathologist using a haematoxylin & eosin (H&E) stained slide.

Secondary aims

To estimate the feasibility of obtaining viable tissue samples at:

* Baseline (sub-cohort 1B)
* PD (Cohort 1)
* Surgery (Cohort 2)

Exploratory aims

* To identify genes/proteins associated with disease progression on targeted therapy (Cohort 1)
* To measure levels of tumour cell-recognising antibodies in patients on targeted therapy (Cohort 1)
* To identify genes/proteins associated with tumour regression (Cohort 2)

ELIGIBILITY:
Inclusion Criteria (Cohort 1):

1. Age >/= 18.
2. Histologically confirmed locally advanced or metastatic NSCLC
3. ECOG performance score 0-2
4. Tier 1 ASCO/AMP NSCLC oncogenic variant identified through routine clinical methods, e.g. EGFR, ALK, ROS1, RET, MET, KRAS, BRAF, HER2, NTRK
5. Planned to commence targeted therapy (any line of therapy)

   o This includes bispecific antibodies (e.g. amivantamab), and antibody-drug conjugates (e.g. trastuzumab-deruxtecan)
6. Regular follow-up and monitoring for cancer recurrence per standard of care planned at the enrolling site
7. Provided written informed consent to participate in the study

Inclusion Criteria (Cohort 2)

1. Age >/= 18.
2. Histologically confirmed stage II/III operable NSCLC
3. Planned to undergo neoadjuvant CPI-based therapy
4. Provided written informed consent to participate in the study

Exclusion Criteria:

• Patient too medically unstable to commit to sampling required for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The Royal Marsden NHS Foundation patients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-06-04 (Actual); Primary Completion 2029-06-01 (Estimated); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
The number of participants with paired samples of blood and viable tissue | 5 years
  The number of participants with paired samples of blood and viable tissue with:
  * Oncogene-addicted metastatic NSCLC commencing new line of targeted therapy at progression (Cohort 1), and
  * Early-stage operable NSCLC undergoing neoadjuvant CPI-based therapy (Cohort 2) Viable tissue is defined by the presence of viable tumour cells. Viable tumour cells are defined by those with well-preserved architectural and cytological features, in line with the latest recommendation from the International Association for the Study of Lung Cancer (IASLC), evaluated by a specialist pulmonary pathologist using a haematoxylin & eosin (H&E) stained slide.

SECONDARY OUTCOMES:
The number of patients with viable tissue samples | 5 years
  The number of patients with viable tissue samples at:
  * Baseline (sub-cohort 1B)
  * PD (Cohort 1)
  * Surgery (Cohort 2)

OTHER OUTCOMES:
Exploratory aims | 5 years
  Exploratory aims
  * The number of genes/proteins associated with disease progression on targeted therapy (Cohort 1)
  * To measure levels of tumour cell-recognising antibodies in patients on targeted therapy (Cohort 1)
  * The number of genes/proteins associated with tumour regression (Cohort 2)

CONTACTS AND LOCATIONS:
Overall Officials: Professor Sanjay Popat, Consultant Medical Oncologist, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- The Royal Marsden NHS Foundation Trust, London, United Kingdom, United Kingdom